CLINICAL TRIAL: NCT03550118
Title: Auto Control of Volume Management for Limb Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Joan Sanders, Professor, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001779
Record Dates: First submitted 2018-05-03; First posted 2018-06-08 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: Prosthetic Socket; Amputee; Adjustable Socket
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (8):
- Aim 2 - Adjustable Socket - Researcher Controls (Experimental): An adjustable socket is tested where researchers control the adjustments. This arm focuses on socket size adjustments while walking.
  Interventions: Device: Adjustable socket
- Aim 3 - Adjustable Socket - Participant Controls (Experimental): An adjustable socket is tested where the study participant controls the adjustments. This arm focuses on socket size adjustments while walking.
  Interventions: Device: Adjustable socket
- Aim 4 - Adjustable Socket - Automatic Controls (Experimental): An adjustable socket is tested where a control system is used to automatically control the adjustments. This arm focuses on socket size adjustments while walking.
  Interventions: Device: Adjustable socket
- Aim 6A - Release/Recovery - Researcher Controls (Experimental): An adjustable socket is tested where researchers control the adjustments. This arm focuses on a socket release and recovery mechanism that allows for full or partial doffing of the socket while seated.
  Interventions: Device: Adjustable socket
- Aim 6B - Release/Recovery - Participant Controls (Experimental): An adjustable socket is tested where the study participant controls the adjustments. This arm focuses on a socket release and recovery mechanism that allows for full or partial doffing of the socket while seated.
  Interventions: Device: Adjustable socket
- Aim 8 - Panel Pull During Resting (Experimental): The purpose of Aim #8 was to determine if vacuum-like action ("panel pull") during resting between periods of activity facilitated limb fluid volume recovery and retention in transtibial prosthesis users. Liner attached to panels.
  Interventions: Device: Adjustable socket
- Aim 9 - Panel Pull During Ambulation (Experimental): Extending from the Aim #8 results, we sought to determine in Aim #9 if "vacuum-like" action during ambulation facilitated limb fluid volume recovery and retention. Vacuum-like action was achieved by quickly pulling the panels and liner (liner attached to panels) radially outward during late stance phase and then moving them back to their original position during early swing.
  Interventions: Device: Adjustable socket
- Aim 10 - Adjustable Socket Out of Lab Testing (Experimental): Participants took the investigational device home in one of three test modes. In the first mode, the panels were in a "locked" flush position, similar to their traditional prosthesis. Participants were not able to adjust the panels in this first mode. The second mode allowed participants to manually make panel adjustments, incrementally enlarging or tightening the panels radially. Lastly, the third mode implemented the automated controller developed in the previous aims. Participants were still able to make manual adjustments to the panel positions but during walks adjustments would also occur automatically. Each mode was tested for a minimum of 1 week.
  Interventions: Device: Adjustable socket

INTERVENTIONS:
Device: Adjustable socket — The adjustable prosthetic socket will be used to test the influence of socket size adjustments during sitting, standing, and walking activities to determine if these strategies can be used to improve socket fit and reduce fluctuations in limb volume.

SUMMARY:
The aim of this research is to create a prosthetic system that will automatically adjust the fit of the socket and create a well-fitting prosthesis for people with leg amputations who experience volume fluctuations when using their prosthesis.

DETAILED DESCRIPTION:
People with lower limb amputations often experience daily changes in the size (volume) of their residual limb. These daily changes can cause a prosthesis to fit poorly. They can also cause limb health problems including skin breakdown and injury to deeper tissues. Prosthetic socket systems that accommodate limb volume changes can help address these issues, but they require users to make adjustments throughout the day.

The objective of this research is to develop and test an automatically-adjusting prosthetic socket system for prosthesis users. The system integrates with a range of adjustable socket technologies, including those that are commercially available. The system allows small size adjustments for both tightening and loosening the socket. In early aims of the study, the prosthesis will be adjusted manually, but can be controlled remotely, eliminating the need to remove the prosthesis or bend down to make adjustments. The system will later be enhanced to automatically change the fit of an adjustable socket at the appropriate times, without distracting the user. We hypothesize that this system will help to maintain consistent limb fluid volume while the prosthesis user is wearing the socket and that socket fit will be improved. The system functions by continuously collecting measurements from sensors within the socket and uses small motors to control adjustable panels in the socket wall.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Unilateral transtibial amputee
* At least 6 months post-amputation
* Wear prosthesis at least 3 hours per day
* Use an elastomeric (i.e. gel) liner
* K3 or higher Medicare Functional Classification Level
* Able to walk continuously with prosthesis for at least 5 minutes at a time, sit, stand, and step up a height of 5.0 cm.
* Residual limb of 9.0 cm or longer
* Experience problems with volume fluctuations that affect their prosthetic socket fit

Exclusion Criteria:

* Participants experiencing skin breakdown on enrollment will be excluded, but can enter after having been free of clinically visually-apparent skin breakdown for two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Sanders, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Bioengineering, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aim 2 - Adjustable Socket - Researcher Controls | Aim 3 - Adjustable Socket - Participant Controls | Aim 4 - Adjustable Socket - Automatic Controls | Aim 6A - Release/Recovery - Researcher Controls | Aim 6B - Release/Recovery - Participant Controls | Aim 8 - Panel Pull During Resting | Aim 9 - Panel Pull During Ambulation | Aim 10 - Adjustable Socket Out of Lab Testing
Started | 15 | 13 | 12 | 13 | 7 | 14 | 12 | 18
Completed | 10 | 12 | 10 | 12 | 6 | 12 | 12 | 12
Not Completed | 5 | 1 | 2 | 1 | 1 | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 2 - Adjustable Socket - Researcher Controls | Aim 3 - Adjustable Socket - Participant Controls | Aim 4 - Adjustable Socket - Automatic Controls | Aim 6A - Release/Recovery - Researcher Controls | Aim 6B - Release/Recovery - Participant Controls | Aim 8 - Panel Pull During Resting | Aim 9 - Panel Pull During Ambulation | Aim 10 - Adjustable Socket Out of Lab Testing | Total
Number analyzed (Participants) | 15 | 13 | 12 | 13 | 7 | 14 | 12 | 18 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 10 | 11 | 6 | 12 | 10 | 14 | 87
  >=65 years | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 4 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 2 | 13
  Male | 13 | 11 | 10 | 11 | 6 | 13 | 11 | 16 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 10
  Not Hispanic or Latino | 13 | 12 | 11 | 12 | 6 | 13 | 11 | 16 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 2 | 13
  White | 10 | 11 | 10 | 11 | 6 | 12 | 10 | 14 | 84
  More than one race | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 12 | 13 | 7 | 14 | 12 | 18 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change in Limb Volume
Description: Limb volume fluctuations will be measured in real-time as socket adjustment strategies are tested. This will be accomplished using a portable bioimpedance device with thin sticky electrodes that are placed on the residual limb. Specifically, the change in limb volume will be assessed from a baseline period where no socket adjustments are made to another period within the same test session where socket adjustments are made.
Time Frame: Change from baseline period (non-adjustment) to test period (adjustment), commonly each 1 hour long and separated by a seated period of approximately 30 minutes.
Population: Change in Limb Volume was monitored only for Arms 2, 6A, 6B, 8 and 9.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 2 - Adjustable Socket - Researcher Controls
Number analyzed (Participants) | 10
Participants
  Experienced limb volume change | 8
  Maintained limb volume | 2

2. Primary Outcome: Change in Limb Movement
Description: Limb movement within the socket will be measured as socket adjustment strategies are tested. It will be used as an indicator of how well the socket is fitting (loose, tight, etc). The measurement will be made using an inductance sensor that is placed in the socket which measures the displacement of a sensor patch on the prosthetic liner. Specifically, the change in limb movement will be assessed from a baseline period where no socket adjustments are made to another period within the same test session where socket adjustments are made.
Time Frame: as for outcome 1
Population: Change in Limb Movement was only measured for Arm 3.
Measure: Median (Full Range); unit: Millimeters
Arm/Group | Aim 3 - Adjustable Socket - Participant Controls
Number analyzed (Participants) | 12
Millimeters
  Sensed Distance, Total Change in Response to Enlargement of Socket Size | 0.01 [-0.13 to 0.11]
  Sensed Distance, Total Change in Response to Reduction of Socket Size | -0.03 [-0.17 to 0.07]

3. Primary Outcome: Change in Limb Volume
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Change in Limb Volume was monitored only for Arms 2, 6A, 6B, 8 and 9.
  Participants were grouped according to their responses to the intervention. The groups "immediate limb volume increase" and "decrease in rate of limb volume loss" presented below are not mutually exclusive. Some participants that experienced immediate limb volume increase were also seen to exhibit a decrease in the rate of limb volume loss.
Measure: Number; unit: participants
Arm/Group | Aim 6A - Release/Recovery - Researcher Controls
Number analyzed (Participants) | 12
participants
  Immediate Limb Volume Increase | 9
  Decrease in rate of limb volume loss | 7

4. Primary Outcome: Change in Limb Volume
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Change in Limb Volume was monitored only for Arms 2, 6A, 6B, 8 and 9.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 6B - Release/Recovery - Participant Controls | Aim 8 - Panel Pull During Resting
Number analyzed (Participants) | 6 | 12
Participants
  Gain in Limb Fluid Volume | 3 | 12
  Loss of Limb Fluid Volume | 3 | 0

5. Primary Outcome: Number of Participants With Increase in Limb Fluid Volume After Panel Pull
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 9 - Panel Pull During Ambulation
Number analyzed (Participants) | 12
Participants | 8

6. Primary Outcome: Integral of Absolute Error to Maintain Set Point
Description: Clinically acceptable socket volume error as measured by an automatically adjusting prosthetic socket attempting to maintain a set socket volume set point, based on sensed distance (measured in mm).
Time Frame: Over 30 minutes of controlled use of the auto-adjusting socket
Measure: Median (Full Range); unit: Millimeters
Arm/Group | Aim 4 - Adjustable Socket - Automatic Controls
Number analyzed (Participants) | 10
Millimeters | 0.003 [0.001 to 0.005]

7. Secondary Outcome: Adjustable Socket Mode Preference
Description: Participants tested the adjustable prosthesis in their home environment in one of three adjustment configurations:
  1. "locked" where panels were kept in position and did not move, similar to their own prosthesis
  2. "manual" where panels were able to be adjusted inward or outward radially, by the participant via a phone app
  3. "automatic" where panels adjusted inward or outward radially as when the participant walked for a sufficiently continuous amount of time. Participants were also able to manual adjust panels as needed in this mode as well.
Time Frame: After 3 weeks of use, where each mode was tested for about 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 10 - Adjustable Socket Out of Lab Testing
Number analyzed (Participants) | 10
Participants
  Preferred Automatic Mode | 5
  Preferred Manual Mode | 5
  Preferred Locked Mode | 0

ADVERSE EVENTS:
Time Frame: Each participant was monitored over the course of their involvement in each Arm's tests, which ranged from same day observations to up to two weeks of out-of-lab testing.
Groups:
- Stress-Sensing Liner: An adjustable socket is tested in addition to a prosthetic liner with embedded stress sensors to measure mechanical stresses as the socket is adjusted.
  Adjustable socket: The adjustable prosthetic socket will be used to test the influence of socket size adjustments during sitting, standing, and walking activities to determine if these strategies can be used to improve socket fit and reduce fluctuations in limb volume.
Arm/Group | Aim 2 - Adjustable Socket - Researcher Controls | Aim 3 - Adjustable Socket - Participant Controls | Aim 4 - Adjustable Socket - Automatic Controls | Stress-Sensing Liner | Aim 6A - Release/Recovery - Researcher Controls | Aim 6B - Release/Recovery - Participant Controls | Aim 8 - Panel Pull During Resting | Aim 9 - Panel Pull During Ambulation | Aim 10 - Adjustable Socket Out of Lab Testing
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/12 | 0/9 | 0/13 | 0/7 | 0/14 | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/12 | 0/9 | 0/13 | 0/7 | 0/14 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/12 | 0/9 | 0/13 | 0/7 | 0/14 | 0/12 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03550118/Prot_SAP_000.pdf